CLINICAL TRIAL: NCT00095862
Title: A Phase 1-2 Study for Stage IV Breast and HER2/Neu Positive Cancers to Evaluate the Safety and Efficacy of a Vaccine Using Whole Cells From the SVBR- 1-GM Cell Line Genetically Engineered To Produce Granulocyte- Macrophage Colony Stimulating Factor
Brief Title: Vaccine Therapy in Treating Patients With HER2/Neu Positive or Negative Stage IV Breast Cancer or Other HER2/Neu Positive Cancers
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wiseman Research Initiatives LLC (Industry)
Responsible Party: Charles L. Wiseman, Wiseman Research Initiatives, LLC
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000393552; WRI-GEV-007
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2011-10

CONDITIONS: Breast Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: recurrent breast cancer; stage IV breast cancer; male breast cancer; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Interferon-alpha; Cyclophosphamide

INTERVENTIONS:
Biological: allogeneic GM-CSF-secreting breast cancer vaccine
Biological: recombinant interferon alfa
Drug: cyclophosphamide

SUMMARY:
RATIONALE: Vaccines made from gene-modified tumor cells may make the body build an immune response to kill tumor cells. Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop tumor cells from dividing so they stop growing or die. Interferon alfa may interfere with the growth of tumor cells. Combining vaccine therapy with cyclophosphamide and interferon alfa may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining vaccine therapy with interferon alfa and cyclophosphamide in treating patients who have stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety, tolerability, and feasibility of vaccine therapy comprising an allogeneic (non-self) tumor cell line transfected with the sargramostim (GM-CSF) gene combined with low-dose interferon alfa and low-dose cyclophosphamide in patients with stage IV breast cancer or other solid tumors.
* Determine the clinical response, time to progression, and survival of patients treated with this regimen.
* Correlate clinical response with immunological response in patients treated with this regimen.

OUTLINE: Patients receive low-dose cyclophosphamide IV once 2-3 days before each tumor vaccine. Patients then receive tumor vaccine comprising HER2/neu-positive allogeneic (non-self) breast cancer cells transfected with the sargramostim (GM-CSF) gene intradermally (ID) on day 1. Patients also receive low-dose interferon alfa ID approximately 48 and 96 hours after each tumor vaccine. Treatment repeats every 2 weeks for 3 vaccinations and then monthly for 3 vaccinations in the absence of disease progression or unacceptable toxicity.

Patients are followed at 2 weeks and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 9-24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer meeting 1 of the following criteria:

  * Recurrent and/or metastatic lesions that are HER2/neu-positive or negative
  * Recurrent or progressive cancer of the lung, ovary, pancreas, prostate, bladder, or other primary site associated with HER2/neu-positive tumor by histochemistry
* Bone-only metastatic breast cancer, cytologically confirmed malignant effusions, histologically confirmed marrow involvement, or other evaluable (but non-measurable) metastatic disease allowed
* Failed prior first-line chemotherapy (e.g., anthracycline- or taxane-based therapy) with or without adjuvant chemotherapy or hormonal therapy
* No curative or reliably effective palliative surgery, radiotherapy, or medical therapy available
* Stable brain metastases allowed provided the following criteria are met*:

  * Previously treated
  * No concurrent requirement for corticosteroids
  * No radiological or clinical deterioration within the past 6 weeks NOTE: *Patients who had recent treatment with gamma knife or intensity-modulated radiotherapy for brain metastases are eligible provided there has been recovery from known or anticipated toxic effects
* Patients with no HLA-A2 allele are eligible
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female or male

Menopausal status

* Not specified

Performance status

* ECOG 0-2

Life expectancy

* At least 4 months

Hematopoietic

* Absolute granulocyte count ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 2 mg/dL
* Alkaline phosphatase ≤ 5 times upper limit of normal (ULN)
* ALT and AST ≤ 2 times ULN

Renal

* BUN ≤ 30 mg/dL
* Creatinine ≤ 2 mg/dL
* ≤ 1 g protein on 24-hour urine collection OR
* ≤ 1+ proteinuria on urinalysis

Cardiovascular

* Hypertension controlled by agents (except beta-blockers) allowed

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No history of anaphylactic reaction to any known or unknown antigen
* No history of clinical hypersensitivity to sargramostim (GM-CSF), interferon, yeast, beef, or to any components used in preparation of study vaccine
* No clinical or laboratory features indicative of AIDS
* No rheumatological, psychiatric, or other clinically progressive major medical problems requiring treatment
* No other malignancy within the past 2 years

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 3 weeks since prior biological therapy, including trastuzumab (Herceptin^®)
* More than 3 weeks since prior immunotherapy
* No concurrent immunotherapy

Chemotherapy

* See Disease Characteristics
* More than 3 weeks since prior chemotherapy (8 weeks for nitrosoureas or mitomycin)
* No concurrent chemotherapy

Endocrine therapy

* See Disease Characteristics
* More than 3 weeks since prior hormonal therapy
* No concurrent hormonal therapy
* No concurrent systemic steroids

  * Concurrent inhalation steroids for respiratory hypersensitivity (e.g., triamcinolone nasal or pulmonary inhalers) allowed

Radiotherapy

* See Disease Characteristics
* More than 3 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery

* More than 3 weeks since prior major surgery with general anesthesia
* No concurrent major surgery

Other

* Recovered from prior therapy
* Patients receiving pamidronate, bisphosphonates, or other supportive measures must continue therapy during study participation
* No concurrent anticoagulants
* No concurrent beta-blockers for control of mild hypertension or other indications

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2004-11

PRIMARY OUTCOMES:
Safety, tolerability, and feasibility
Clinical response
Time to progression
Survival
Correlation of clinical response with immunological response

CONTACTS AND LOCATIONS:
Overall Officials: Charles L. Wiseman, MD, FACP, Study Chair
Locations (3):
- United States (3):
  - Glendale Memorial Hospital Comprehensive Cancer Center, Glendale, California
  - Hollywood Presbyterian Medical Center, Los Angeles, California
  - Los Angeles, California

REFERENCES:
- [Derived] Lacher MD, Bauer G, Fury B, Graeve S, Fledderman EL, Petrie TD, Coleal-Bergum DP, Hackett T, Perotti NH, Kong YY, Kwok WW, Wagner JP, Wiseman CL, Williams WV. SV-BR-1-GM, a Clinically Effective GM-CSF-Secreting Breast Cancer Cell Line, Expresses an Immune Signature and Directly Activates CD4+ T Lymphocytes. Front Immunol. 2018 May 15;9:776. doi: 10.3389/fimmu.2018.00776. eCollection 2018. PMID 29867922